CLINICAL TRIAL: NCT05790551
Title: Development of a Telehealth Medication-assisted Treatment (MAT) System for Patients With Opioid Use Disorder (OUD)
Brief Title: Suboxone Dispenser for OUD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was discontinued at the primary site due to change in site management.
Sponsor: Addinex Technologies, Inc. (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R43CE003533 (NIH)
Record Dates: First submitted 2023-02-24; First posted 2023-03-30 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder; Opioid Withdrawal
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): Patients in this arm will undergo standard at-home OUD treatment (n = 5/group) over 14-days.
  Interventions: Device: Addinex
- Active - App (Experimental): Patients in this arm will undergo standard at-home OUD treatment in combination with the Addinex dispenser and app (n = 5/group) over 14-days.
  Interventions: Device: Addinex

INTERVENTIONS:
Device: Addinex — Medication dispensing system for Suboxone

SUMMARY:
The goal of this study is to evaluate the usability and acceptability of the Addinex system with patients receiving Suboxone in OUD treatment. The main questions it aims to answer are:

* Are patients more likely to stay on their medication?
* Is the risk of diversion being reduced?
* How is the usability of the Addinex system for doctors and patients?

DETAILED DESCRIPTION:
Prescription opioids remain a popular drug class with 142 million (M) opioid prescriptions written in 2020. In that same year, 9.5M people aged 12 or older misused opioids representing 3.3% of that population and overdose deaths from opioids rose to 70,029, an increase of 37% (which has since increased to 82,310 in 2021). The COVID-19 pandemic has exposed many vulnerabilities in the treatment of patients with OUD. Of patients prescribed opioids, between 3-10% will later develop opioid use disorder (OUD). Given that prescription opioids remain the dominant route through which OUD begins, reducing their abuse and diversion can translate over time into reduced deaths.

Many patients with OUD are treated by a combination of buprenorphine with counseling and behavioral therapies, also known as Medication Assisted Treatment (MAT). Although buprenorphine is less addictive than opioids or other treatments (e.g., methadone), it is not invulnerable to abuse or diversion. There is therefore a significant opportunity for the development of new technologies aimed at remotely treating OUD, and preventing drug misuse, abuse, and diversion. Although several secure dispenser technologies are under development, there remains a critical need for a comprehensive solution that prevents and/or treats addiction, tracks usage, collects data, and eliminates excess medication, while also remaining modular and cost effective enough to be widely accessible.

Addinex Technologies, Inc. is developing the only solution that combines: 1) a patented, secure, low-cost and modular medication-dispenser which controls medication access and encourages convenient and safe unused medication disposal, combined with 2) companion mobile patient app and physician/pharmacist web-based software that features interactive modules and surveys to improve patient education and engagement, caregiver monitoring, and teletherapy to facilitate patient-provider interactions.

Addinex will conduct a feasibility and acceptability study for its app-based and text-based system across patients (n = 60) undergoing OUD treatment. Successful completion of these aims will provide critical insights to further optimize the Addinex system and to guide the design of a larger, randomized controlled trial to demonstrate its efficacy and cost effectiveness.

This study will be the springboard for the development of a system that is cost efficient, widely accessible, and user-friendly, with the aim of increasing adherence, decreasing treatment time, decreasing the misuse of medication, increasing treatment retention, and reducing relapses in OUD treatment for the many who are suffering.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 18 years old at admission of study
* Primary or secondary diagnosis of opioid use disorder (DSM-5; APA, 2013) diagnosis by clinician
* Prospective patients have to select 'Yes' they are interested in Yale-approved research studies while enrolled at Aware Recovery Care and that researchers can contact them about research projects

Exclusion Criteria:

* Meets criterion of DSM-V (APA, 2013) for bi-polar, schizophrenia, or psychiatric disorders
* Unable to read and understand English at 5th grade level
* Unable to complete the study because of anticipated incarceration or move
* Life threatening or unstable medical problems
* Current suicide or homicide risk
* Anticipated/current pregnancy, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Drug Test for Opioid Use Disorder (Quest 12-Panel Drug Screen) | Up to two weeks
  Urine analysis will be completed on a biweekly basis for the research study

SECONDARY OUTCOMES:
PROMIS Self-Efficacy Scale | Up to two weeks
  Evaluation of participants' self-efficacy toward change over the course of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Greenwich Hospital, Greenwich, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No